CLINICAL TRIAL: NCT00830167
Title: Randomized, Double-Blind, Multicenter, Placebo-Controlled Study To Evaluate Efficacy And Safety Of Pregabalin（CI-1008）In The Treatment Of Fibromyalgia
Brief Title: Randomized, Double-Blind, Placebo-Controlled Study Of Pregabalin In Patients With Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081208
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2012-04

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Placebo — Dosage: placebo, oral administration, Treatment duration: 15 weeks (3-week titration and 12-week fixed dose)
  Arms: Placebo
Drug: Pregabalin — Dosage: 300 or 450 mg/day (150 or 225 mg bid), oral administration, Treatment duration: 15 weeks (3-week titration and 12-week fixed dose)
  Arms: Pregabalin

SUMMARY:
This study, will compare pregabalin with placebo for the duration of 15 weeks to evaluate the efficacy and safety of pregabalin in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* ACR criteria for fibromyalgia
* A score of more or equal to 40 mm on the Pain VAS
* An average score more or equal to 4 on 4 daily pain diaries

Exclusion Criteria:

* Patients with other severe pain conditions
* Patients with severe depression
* Patients taking excluded medications
* Patients with suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- Japan (35):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Ichihara-shi, Chiba
  - Pfizer Investigational Site, Yotukaidou, Chiba
  - Pfizer Investigational Site, Matuyama-si, Ehime
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Iiduka, Fukuoka
  - Pfizer Investigational Site, Kitakyushu, Fukuoka
  - Pfizer Investigational Site, Takasaki, Gunma
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Kobe, Hyōgo
  - Pfizer Investigational Site, Mito, Ibaraki
  - Pfizer Investigational Site, Morioka, Iwate
  - Pfizer Investigational Site, Sagamihara-shi, Kanagawa
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Koushi, Kumamoto
  - Pfizer Investigational Site, Tsu, Mie-ken
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Hiki-gun, Saitama
  - Pfizer Investigational Site, Saitama, Saitama
  - Pfizer Investigational Site, Saitama-shi, Saitama
  - Pfizer Investigational Site, Aoi-ku, Shizuoka
  - Pfizer Investigational Site, Shimotsuga-gun, Tochigi
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Chiyoda-ku, Tokyo
  - Pfizer Investigational Site, Chuou-Ku, Tokyo
  - Pfizer Investigational Site, Itabashi-Ku, Tokyo
  - Pfizer Investigational Site, Setagaya City, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Shinagawa-Ku, Tokyo
  - Pfizer Investigational Site, Toyama, Toyama
  - Pfizer Investigational Site, Nagano
  - Pfizer Investigational Site, Osaka
  - Pfizer Investigational Site, Ōita
  - Pfizer Investigational Site, Tokushima
  - Pfizer Investigational Site, Yokohama

REFERENCES:
- [Derived] Clair A, Emir B. The safety and efficacy of pregabalin for treating subjects with fibromyalgia and moderate or severe baseline widespread pain. Curr Med Res Opin. 2016;32(3):601-9. doi: 10.1185/03007995.2015.1134463. Epub 2016 Jan 27. PMID 26694975
- [Derived] Ohta H, Oka H, Usui C, Ohkura M, Suzuki M, Nishioka K. A randomized, double-blind, multicenter, placebo-controlled phase III trial to evaluate the efficacy and safety of pregabalin in Japanese patients with fibromyalgia. Arthritis Res Ther. 2012 Oct 12;14(5):R217. doi: 10.1186/ar4056. PMID 23062189
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081208&StudyName=Randomized%2C%20Double-Blind%2C%20Placebo-Controlled%20Study%20Of%20Pregabalin%20In%20Patients%20With%20Fibromyalgia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were administered placebo tablet in single blind manner and evaluated for the inclusion/exclusion criteria during the 1-week screening phase. Participants who demonstrated a high response to placebo, i.e., <=30% decrease on the VAS, were discontinued from the study at the end of the screening phase.
Groups:
- Placebo: Placebo was administered twice a day for 15 weeks.
- Pregabalin: Pregabalin was administered twice a day at the starting dose of 150 mg/day in the first week and escalated to 300 mg/day at the end of Week 1. Pregabalin dose was titrated to 450 mg/day at the end of Week 2 based on the participant's individual response and tolerability to pregabalin. Treatment period was 15 weeks that consisted of 3-week dose optimization phase and 12-week fixed dose phase.
Period: Overall Study
Arm/Group | Placebo | Pregabalin
Started | 248 (Treated) | 250 (Treated)
Completed | 208 | 207
Not Completed | 40 | 43
Not completed — Lack of Efficacy | 26 | 10
Not completed — Adverse Event | 8 | 24
Not completed — Not meeting entrance criteria | 2 | 5
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin | Total
Number analyzed (Participants) | 248 | 250 | 498
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0
  Between 18 years and 44 years | 104 | 101 | 205
  Between 45 years and 64 years | 123 | 125 | 248
  >=65 years | 21 | 24 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 226 | 443
  Male | 31 | 24 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for Numerical Rating Scale (NRS) Pain Scores at Endpoint-LOCF (Last Observation Carried Forward) Relative to Baseline
Description: Change from baseline in mean NRS-Pain scores at endpoint-LOCF. Daily pain scores were assessed on an 11-point numerical rating scale <(NRS)-Pain> ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 15 or study discontinuation
Population: The full analysis set (FAS) consisted of all randomized participants who received at least 1 dose of study medication and had at least 1 postbaseline pain score on study medication. Last observation carried forward (LOCF) method was used.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -1.03 (0.12) | -1.48 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; The null hypothesis was to assume that there was no difference between the pregabalin and placebo groups. The alternative was that the pregabalin group was superior to the placebo group; Test type: Superiority or Other; p = 0.0046, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025. Actual significance level was calculated based on O'Brien-Fleming type alpha spending function of Lan and DeMets (1983); Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.78 to -0.11], Standard Error of Mean 0.17

2. Secondary Outcome: Percentage of Participants Who Was Categorized as "Improved (Very Much Improved, Much Improved, or a Minimally Improved)" According to the Patient Global Impressions of Change (PGIC)
Description: PGIC was defined as participant rated instrument to measure participant's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse). Change was defined as a score of 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse) , 6 (much worse) or 7 (very much worse) on the scale.
Time Frame: Week 15 or study discontinuation
Population: The full analysis set (FAS) consisted of all randomized participants who received at least 1 dose of study medication and had at least 1 postbaseline pain score on study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 247 | 249
Percentage of participants | 62.1 | 70.0
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; The null hypothesis was to assume that there was no difference between the pregabalin and placebo groups. The alternative was that there was a difference between the pregabalin and the placebo groups; Test type: Superiority or Other; p = 0.0078, Chi-squared — The analysis was conducted using 2-sided test with the significance level of 0.05

3. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale at Endpoint- Sleep Disturbance
Description: MOS: participant-rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Sleep Disturbance subscales rated 1 (all the time) to 6 (none of the time). Scores are transformed (actual raw score minus lowest possible score) divided by possible raw score range multiplied by 100; total score range = 0 to 100. A higher score indicates greater intensity of sleep disturbance. Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 247 | 249
Scores on a scale | -8.13 (1.31) | -17.62 (1.31)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -9.48, 95% CI 2-sided [-13.12 to -5.85], Standard Error of Mean 1.85

4. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale at Endpoint- Snoring
Description: MOS: participant-rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Snoring subscales rated 1 (all the time) to 6 (none of the time). Scores are transformed (actual raw score minus lowest possible score) divided by possible raw score range multiplied by 100; total score range = 0 to 100. A higher score indicates greater intensity of snoring. Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 247 | 249
Scores on a scale | -1.61 (1.33) | 3.37 (1.33)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9958, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = 4.98, 95% CI 2-sided [1.29 to 8.68], Standard Error of Mean 1.88

5. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale at Endpoint- Awaken Short of Breath or With a Headache
Description: MOS: participant-rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Awaken Short of Breath or With a Headache subscales rated 1 (all the time) to 6 (none of the time). Scores are transformed (actual raw score minus lowest possible score) divided by possible raw score range multiplied by 100; total score range = 0 to 100. A higher score indicates greater intensity of the symptom. Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 247 | 249
Scores on a scale | -3.02 (1.36) | -8.01 (1.36)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0049, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -4.99, 95% CI 2-sided [-8.77 to -1.21], Standard Error of Mean 1.92

6. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale at Endpoint- Quantity of Sleep
Description: MOS: participant-rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Quantity of Sleep subscales rated 0 to 24 (number of hours slept). A higher score indicates greater quantity of sleep. Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 247 | 249
Scores on a scale | 0.17 (0.06) | 0.46 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0007, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [0.11 to 0.47], Standard Error of Mean 0.09

7. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale at Endpoint- Sleep Adequacy
Description: MOS: participant-rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Sleep Adequacy subscales rated 1 (all the time) to 6 (none of the time). Scores are transformed (actual raw score minus lowest possible score) divided by possible raw score range multiplied by 100; total score range = 0 to 100. A higher score indicates greater intensity of sleep adequacy. Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 247 | 249
Scores on a scale | 8.02 (1.41) | 15.50 (1.40)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = 7.48, 95% CI 2-sided [3.58 to 11.38], Standard Error of Mean 1.99

8. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale at Endpoint- Somnolence
Description: MOS: participant-rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Somnolence subscales rated 1 (all the time) to 6 (none of the time). Scores are transformed (actual raw score minus lowest possible score) divided by possible raw score range multiplied by 100; total score range = 0 to 100. A higher score indicates greater intensity of somnolence. Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 247 | 249
Scores on a scale | -4.66 (1.29) | 6.65 (1.28)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.0000, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = 11.31, 95% CI 2-sided [7.74 to 14.87], Standard Error of Mean 1.82

9. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale at Endpoint- Overall Sleep Problems Index
Description: MOS: participant-rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Overall Sleep Problems Index subscales rated 1 (all the time) to 6 (none of the time). Scores are transformed (actual raw score minus lowest possible score) divided by possible raw score range multiplied by 100; total score range = 0 to 100. A higher score indicates greater intensity of overall sleep problems. Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 247 | 249
Scores on a scale | -7.07 (0.96) | -10.06 (0.95)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0137, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -2.99, 95% CI 2-sided [-5.65 to -0.33], Standard Error of Mean 1.35

10. Secondary Outcome: Medical Outcomes Study (MOS) Sleep Scale - Number of Participants With Optimal Sleep at Endpoint
Description: MOS-Sleep is a patient-rated questionnaire to assess sleep quality and quantity. Optimal sleep component is derived from Sleep Quantity average hours of sleep each night during the past 4 weeks. Optimal sleep was defined as sleep quantity of 7 or 8 hours per night.
Time Frame: Week 15 or study discontinuation
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 247 | 249
Participants | 53 | 71
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0687, Regression, Logistic — The analysis was conducted using 1-sided test with the significance level of 0.025; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.90 to 2.35]

11. Secondary Outcome: Change From Baseline in Sleep Quality Score at Endpoint
Description: Change: Mean sleep quality score at endpoint minus mean at baseline. Sleep quality scores range from 0-10 with higher scores indicating decreased sleep quality.
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -0.79 (0.12) | -1.52 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-1.06 to -0.40], Standard Error of Mean 0.17

12. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) at Endpoint - Total Scores
Description: FIQ is a 20-item patient-reported outcome instrument designed to assess health status, progress, and outcomes in patients with fibromyalgia (10 subscales; 11 questions). Scores range from 0 to 100 with higher scores indicating more impairment. Change = mean FIQ scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -7.26 (1.08) | -10.59 (1.07)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0144, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -3.33, 95% CI 2-sided [-6.31 to -0.35], Standard Error of Mean 1.52

13. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) at Endpoint - Physical Function
Description: as for outcome 12
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -0.19 (0.11) | -0.47 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0376, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.59 to 0.03], Standard Error of Mean 0.16

14. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) at Endpoint - Feel Good
Description: as for outcome 12
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -0.82 (0.17) | -1.45 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0052, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.12 to -0.15], Standard Error of Mean 0.25

15. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) at Endpoint - Work Miss
Description: as for outcome 12
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -0.30 (0.15) | -0.31 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4768, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.42 to 0.40], Standard Error of Mean 0.21

16. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) at Endpoint - Housework
Description: as for outcome 12
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -1.00 (0.15) | -1.32 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0729, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.74 to 0.11], Standard Error of Mean 0.21

17. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) at Endpoint - Pain
Description: as for outcome 12
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -1.06 (0.15) | -1.46 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0238, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.81 to 0.00], Standard Error of Mean 0.21

18. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) at Endpoint - Tiredness
Description: as for outcome 12
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -0.94 (0.14) | -1.43 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0075, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.89 to -0.10], Standard Error of Mean 0.20

19. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) at Endpoint - Morning
Description: as for outcome 12
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -0.97 (0.15) | -1.56 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0023, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-1.01 to -0.18], Standard Error of Mean 0.21

20. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) at Endpoint - Stiffness
Description: as for outcome 12
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -0.90 (0.15) | -1.05 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2568, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.57 to 0.29], Standard Error of Mean 0.22

21. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) at Endpoint - Anxious
Description: as for outcome 12
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -0.64 (0.16) | -0.92 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1011, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.72 to 0.15], Standard Error of Mean 0.22

22. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) at Endpoint - Depression
Description: as for outcome 12
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -0.51 (0.14) | -0.55 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4165, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.44 to 0.35], Standard Error of Mean 0.20

23. Secondary Outcome: Change From Baseline in Analysis of SF-36 Health Survey Results at Endpoint- Physical Functioning
Description: Subject-rated measure of health status comprised of 36 items: 8 subscale scores (physical functioning, role limitations-physical, bodily pain, general health perceptions, vitality, social functioning, role limitations-emotional, and mental health. Subscale scores range: 0-100. Higher subscale scores = better health status. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | 4.72 (0.93) | 9.01 (0.93)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0006, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = 4.29, 95% CI 2-sided [1.70 to 6.88], Standard Error of Mean 1.32

24. Secondary Outcome: Change From Baseline in Analysis of SF-36 Health Survey Results at Endpoint- Role Limitations-Physical
Description: as for outcome 23
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | 8.36 (1.30) | 10.04 (1.30)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1805, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = 1.68, 95% CI 2-sided [-1.93 to 5.29], Standard Error of Mean 1.84

25. Secondary Outcome: Change From Baseline in Analysis of SF-36 Health Survey Results at Endpoint- Bodily Pain
Description: as for outcome 23
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | 9.50 (1.06) | 11.65 (1.06)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0770, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = 2.15, 95% CI 2-sided [-0.81 to 5.10], Standard Error of Mean 1.50

26. Secondary Outcome: Change From Baseline in Analysis of SF-36 Health Survey Results at Endpoint- General Health Perception
Description: as for outcome 23
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | 2.83 (0.85) | 4.66 (0.85)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0648, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = 1.83, 95% CI 2-sided [-0.54 to 4.19], Standard Error of Mean 1.20

27. Secondary Outcome: Change From Baseline in Analysis of SF-36 Health Survey Results at Endpoint- Social Functioning
Description: as for outcome 23
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | 6.84 (1.38) | 8.43 (1.37)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2068, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = 1.59, 95% CI 2-sided [-2.23 to 5.41], Standard Error of Mean 1.94

28. Secondary Outcome: Change From Baseline in Analysis of SF-36 Health Survey Results at Endpoint- Role Limitations-Emotional
Description: as for outcome 23
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | 3.50 (1.36) | 3.27 (1.35)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5480, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-4.00 to 3.54], Standard Error of Mean 1.92

29. Secondary Outcome: Change From Baseline in Analysis of SF-36 Health Survey Results at Endpoint- Vitality
Description: as for outcome 23
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | 5.12 (1.22) | 9.53 (1.21)
Statistical Analysis 1: Comparison: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0052, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = 4.42, 95% CI 2-sided [1.04 to 7.80], Standard Error of Mean 1.72

30. Secondary Outcome: Change From Baseline in Analysis of SF-36 Health Survey Results at Endpoint- Mental Health
Description: as for outcome 23
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | 3.33 (0.98) | 5.97 (0.98)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0287, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = 2.64, 95% CI 2-sided [-0.08 to 5.37], Standard Error of Mean 1.39

31. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) - Anxiety
Description: Change: Mean HADS score at observation minus Mean at baseline. HADS anxiety and depression subscale scores range from 0 to 21, with higher scores indicating greater severity of the subscale condition.
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 247 | 249
Scores on a scale | -0.09 (0.18) | -0.57 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0262, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.97 to 0.01], Standard Error of Mean 0.25

32. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) - Depression
Description: as for outcome 31
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 247 | 249
Scores on a scale | 0.00 (0.20) | -0.29 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1561, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.83 to 0.27], Standard Error of Mean 0.28

33. Secondary Outcome: Change From Baseline in Pain Visual Analog Scale (Pain VAS) Score at Endpoint
Description: The pain VAS is a horizontal line; 100 mm in length, self-administered by the patient to rate pain from 0 (no pain) to 100 (worst possible pain). The score indicates the pain intensity during the past 1 week before a visit. Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 15 or study discontinuation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 248 | 250
Scores on a scale | -14.11 (1.45) | -20.30 (1.44)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0013, ANCOVA — The analysis was conducted using 1-sided test with the significance level of 0.025; Mean Difference (Final Values) = -6.19, 95% CI 2-sided [-10.20 to -2.18], Standard Error of Mean 2.04

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/248 | 1/250
Other Adverse Events (participants affected / at risk) | 113/248 | 195/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=248) | Pregabalin (N=250)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=248) | Pregabalin (N=250)
Vision blurred (Eye disorders) | 3 | 13
Constipation (Gastrointestinal disorders) | 17 | 36
Feeling abnormal (General disorders) | 3 | 20
Oedema peripheral (General disorders) | 3 | 18
Nasopharyngitis (Infections and infestations) | 45 | 45
Weight increased (Investigations) | 9 | 39
Dizziness (Nervous system disorders) | 15 | 74
Headache (Nervous system disorders) | 15 | 15
Somnolence (Nervous system disorders) | 45 | 116

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.